CLINICAL TRIAL: NCT06786143
Title: The Effect of Esmadem Education Model on Spiritual Coping, Tolerance and Depression of High-Risk Pregnant Women
Brief Title: Esmadem Education Model on High-Risk Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Mine Gokduman Keles, PhD midwife, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 08.01.2025/01/25decision no
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Risky Pregnancies
Keywords: risky pregnancies; Education; Spiritual; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention)
- INTERVENTION 1 (Experimental)
  Interventions: Behavioral: Esmadem Education Model

INTERVENTIONS:
Behavioral: Esmadem Education Model — Application Application of the Research The implementation of the research was done in 3 steps.
  Step 1: In the first stage of the research, after the risky pregnant women who come to the polyclinic are informed about the study, the participants who agree to participate and meet the criteria for inclusion in the research will be determined by randomization. After the pregnant women assigned to the training or control group sign the voluntary consent form and their consent is obtained, Personal InformationForm, Mishel Uncertainty in Illness Scale Depression-Anxiety-Stress Scale Depression-Anxiety-Stress Scale (DASÖ-21) scales will be applied. After the first interviews, the study group will be informed about the sessions and the training will start via zoom.
  In educational sciences, since the number of groups is between 2-20 people in the acquisition of target behaviors at the conceptual level, two training groups will be created and 15 pregnant women will be in the first group, 15 preg
  Arms: INTERVENTION 1

SUMMARY:
Pregnancy is a normal and natural process in a woman's life. During this process, anatomical, physiological, biochemical and emotional changes are observed. During pregnancy, sometimes risk situations arise from the mother, sometimes from the fetus. the scope of prenatal care is high today, the main focus is on the physical aspects of care and medical measures. Midwives who provide holistic care should also address spiritual care. Therefore, the esmadem education model will be conducted to examine the effect of the spiritual coping, tolerance and depression of risky pregnancies.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women aged 18-45 ,In the second trimester, Primiparous, Have sufficient communication skills, Literate, Can read and understand Turkish, Agree to participate in the research Continuing pregnancy school Having a risky pregnancy diagnosis according to the criteria in the Ministry of Health Pregnancy Risk Assessment Form and having been diagnosed as a risky pregnancy by a physician

Exclusion Criteria:

* Having any mental illness

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Religious Coping Scale | aseline and 3 months.
Michel Uncertainty Scale in Illness-Community Form, | aseline and 3 months.
Depression-Anxiety-Stress Scale | aseline and 3 months.